CLINICAL TRIAL: NCT06504693
Title: Iron Status in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Iron Status in Children With ADHD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Safwat Finiar Fanous, Doctor, Assiut University
Other Study IDs: Iron status in ADHD
Record Dates: First submitted 2024-07-09; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC — diagnostic tests for iron status
  Other Names: Serum ferritin level; Serum iron level

SUMMARY:
Evaluation of the status of iron deficiency in children with attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is one of the most prevalent neurodevelopmental disorders, affecting ~5-8% of children worldwide. For about 60% children with ADHD, the symptoms persist into adulthood. Individuals with ADHD have poorer educational and social outcomes, increased injury incidences during daily activities and an elevated risk of developing more severe mental disorders.

Attention deficit/hyperactivity disorder (ADHD) is a neurodevelopmental disorder defined by persistent, impairing and developmentally inappropriate inattentive/disorganized and/or hyperactive/impulsive behaviors that lie at the far end of a normally distributed continuum.

Dopamine is one of the key neurotransmitters in the brain. Besides its regulatory role in motor and limbic functions, dopamine also regulates cognition, attention, and reward, each of which is impaired in ADHD. The nigrostriatal dopamine pathway is involved in motor control, while the mesolimbic dopamine pathway is involved in motivation and reinforcement learning. The mesocortical dopamine pathway originating in the ventral tegmental area (VTA) and projecting to the prefrontal cortex (PFC) plays a role in cognitive functioning.

Brain iron homeostasis may be important in the pathophysiology of ADHD because iron is a cofactor of the rate-limiting enzyme tyrosine hydroxylase, which is required for dopamine synthesis in the metabolism of dopamine and the hypodopaminergic state of the brain in ADHD results in the symptoms of the disorder. Moreover, iron is colocalized with dopamine in the brain of children with ADHD.

In children, iron deficiency can therefore lead to delayed cognitive, motor, attention and memory deficits, visual and auditory deficits, decreased school performance, and/or behavioral disorders, some with persistent long-term effects.

WHO defines anemia in a population as a mild, moderate, or severe public health problem if its prevalence is 5-20%, 20-40%, or >40%, respectively. Most of the WHO countries have a moderate-to-severe public health problem with anemia, i.e., over 20% of women and young children are affected. In developing countries, diets with poor iron bioavailability are the primary cause of iron deficiency anemia.

There is a high demand for dietary iron during infancy and preschool years to support physical growth, rapid brain development, and early learning capacity.Prompt identification and treatment of anemia leads to overall improvement of population health outcomes, improved physical exercise performance, and well-being that results in enhanced economic productivity.

ELIGIBILITY:
Inclusion Criteria:

* All children above 4 years and under 12 years old diagnosed with attention deficit hyperactivity disorder (ADHD) according to DSM-V criteria.
* Not receiving iron therapy

Exclusion Criteria:

* Children under 4 years old
* Above 12 years old
* Not diagnosed attention deficit hyperactivity disorder(ADHD)
* Any other associated neurological disorder

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children above 4 years and under 12 years old diagnosed with attention deficit hyperactivity disorder (ADHD)
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Iron status in children with attention deficit hyperactivity disorder | Baseline
  To determine number of patients with ADHD who have associated iron deficiency

REFERENCES:
- [Background] Mantadakis E, Chatzimichael E, Zikidou P. Iron Deficiency Anemia in Children Residing in High and Low-Income Countries: Risk Factors, Prevention, Diagnosis and Therapy. Mediterr J Hematol Infect Dis. 2020 Jul 1;12(1):e2020041. doi: 10.4084/MJHID.2020.041. eCollection 2020. PMID 32670519
- See also: Related Info — http://doi.org/10.1038/s41390-020-0907-5
- See also: Related Info — http://doi.org/10.1007/s00787-021-01871-x
- See also: Related Info — http://doi.org/10.1038/s41398-023-02536-w
- See also: Related Info — http://doi.org/10.1007/s00431-020-03597-5
- See also: Related Info — http://doi.org/10.1007/978-3-030-42825-9_33-1